CLINICAL TRIAL: NCT01981772
Title: Anesthetic Efficacy of 4% Buffered Lidocaine in Emergency Patients With Facial Swelling.
Brief Title: Efficacy of Buffered Lidocaine in Patients With Facial Swelling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Melissa Drum, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012H0437
Record Dates: First submitted 2013-07-31; First posted 2013-11-13 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Orofacial Swelling
MeSH Terms: interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- buffered lidocaine (Experimental): administration of 4% buffered lidocaine with 1:100,000 epinephrine
  Interventions: Drug: 4% buffered lidocaine with 1:100,000 epinephrine
- nonbuffered lidocaine (Active Comparator): administration of 4% lidocaine with 1:100,000 epinephrine
  Interventions: Drug: 4% lidocaine with 1:100,000 epinephrine

INTERVENTIONS:
Drug: 4% lidocaine with 1:100,000 epinephrine — see arm/group description
  Arms: nonbuffered lidocaine
Drug: 4% buffered lidocaine with 1:100,000 epinephrine — see arm/group description
  Arms: buffered lidocaine

SUMMARY:
The purpose of this study is to determine the clinical efficacy of a buffered 4% lidocaine solution for incision and drainage. Ninety patients will be examined clinically to determine a diagnosis of cellulitis or fluctuance. The diagnosis will be confirmed by incision and drainage. Patients will receive either 3.6 ml 4% lidocaine with 1:100,000 epinephrine or 3.6 ml 4% lidocaine with 1:100,000 epinephrine buffered with 8.4% sodium bicarbonate. Patients will rate pain prior to and throughout the procedure.

DETAILED DESCRIPTION:
Incision and drainage of swellings is painful and anesthetic failure is common. One reason may be related to the lowered pH of inflamed tissue reducing the amount of the base form of anesthetic. A buffered anesthetic solution may result in more effective anesthesia than a non-buffered solution.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* in good health (ASA classification I or II)
* able to give informed consent
* necrotic tooth with associated facial swelling

Exclusion Criteria:

* allergies to local anesthetics or sulfites
* history of significant medical problems (ASA classification III or greater)
* pregnancy
* inability to give informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Drum, DDS, MS, Principal Investigator — The Ohio State University College of Dentistry
Locations (1):
- The Ohio State University College of Dentistry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adhikari S, Blaivas M, Lander L. Comparison of bedside ultrasound and panorex radiography in the diagnosis of a dental abscess in the ED. Am J Emerg Med. 2011 Sep;29(7):790-5. doi: 10.1016/j.ajem.2010.03.005. Epub 2010 May 1. PMID 20825898
- [Background] Singer AJ, Richman PB, Kowalska A, Thode HC Jr. Comparison of patient and practitioner assessments of pain from commonly performed emergency department procedures. Ann Emerg Med. 1999 Jun;33(6):652-8. PMID 10339680
- [Background] Strichartz GR. Novel ideas of local anaesthetic actions on various ion channels to ameliorate postoperative pain. Br J Anaesth. 2008 Jul;101(1):45-7. doi: 10.1093/bja/aen101. Epub 2008 May 16. PMID 18487246
- [Background] Cohen JS, Reader A, Fertel R, Beck M, Meyers WJ. A radioimmunoassay determination of the concentrations of prostaglandins E2 and F2alpha in painful and asymptomatic human dental pulps. J Endod. 1985 Aug;11(8):330-5. doi: 10.1016/s0099-2399(85)80039-x. No abstract available. PMID 3863874
- [Background] Isett J, Reader A, Gallatin E, Beck M, Padgett D. Effect of an intraosseous injection of depo-medrol on pulpal concentrations of PGE2 and IL-8 in untreated irreversible pulpitis. J Endod. 2003 Apr;29(4):268-71. doi: 10.1097/00004770-200304000-00010. PMID 12701778
- [Background] Wells JE, Bingham V, Rowland KC, Hatton J. Expression of Nav1.9 channels in human dental pulp and trigeminal ganglion. J Endod. 2007 Oct;33(10):1172-6. doi: 10.1016/j.joen.2007.05.023. Epub 2007 Aug 27. PMID 17889684
- [Background] Luo S, Perry GM, Levinson SR, Henry MA. Nav1.7 expression is increased in painful human dental pulp. Mol Pain. 2008 Apr 21;4:16. doi: 10.1186/1744-8069-4-16. PMID 18426592
- [Background] Warren CA, Mok L, Gordon S, Fouad AF, Gold MS. Quantification of neural protein in extirpated tooth pulp. J Endod. 2008 Jan;34(1):7-10. doi: 10.1016/j.joen.2007.09.014. Epub 2007 Nov 26. PMID 18155483
- [Background] Owatz CB, Khan AA, Schindler WG, Schwartz SA, Keiser K, Hargreaves KM. The incidence of mechanical allodynia in patients with irreversible pulpitis. J Endod. 2007 May;33(5):552-6. doi: 10.1016/j.joen.2007.01.023. Epub 2007 Mar 6. PMID 17437870
- [Background] Modaresi J, Dianat O, Soluti A. Effect of pulp inflammation on nerve impulse quality with or without anesthesia. J Endod. 2008 Apr;34(4):438-41. doi: 10.1016/j.joen.2008.01.014. Epub 2008 Mar 4. PMID 18358891
- [Background] Roy ML, Narahashi T. Differential properties of tetrodotoxin-sensitive and tetrodotoxin-resistant sodium channels in rat dorsal root ganglion neurons. J Neurosci. 1992 Jun;12(6):2104-11. doi: 10.1523/JNEUROSCI.12-06-02104.1992. PMID 1318956
- [Background] Bartfield JM, Homer PJ, Ford DT, Sternklar P. Buffered lidocaine as a local anesthetic: an investigation of shelf life. Ann Emerg Med. 1992 Jan;21(1):16-9. doi: 10.1016/s0196-0644(05)82230-9. PMID 1539881
- [Background] Zahl K, Jordan A, McGroarty J, Sorensen B, Gotta AW. Peribulbar anesthesia. Effect of bicarbonate on mixtures of lidocaine, bupivacaine, and hyaluronidase with or without epinephrine. Ophthalmology. 1991 Feb;98(2):239-42. doi: 10.1016/s0161-6420(91)32311-x. PMID 2008283
- [Background] Sinnott CJ, Garfield JM, Thalhammer JG, Strichartz GR. Addition of sodium bicarbonate to lidocaine decreases the duration of peripheral nerve block in the rat. Anesthesiology. 2000 Oct;93(4):1045-52. doi: 10.1097/00000542-200010000-00028. PMID 11020760
- [Background] Richtsmeier AJ, Hatcher JW. Buffered lidocaine for skin infiltration prior to hemodialysis. J Pain Symptom Manage. 1995 Apr;10(3):198-203. doi: 10.1016/0885-3924(94)00124-4. PMID 7629414
- [Background] Burns CA, Ferris G, Feng C, Cooper JZ, Brown MD. Decreasing the pain of local anesthesia: a prospective, double-blind comparison of buffered, premixed 1% lidocaine with epinephrine versus 1% lidocaine freshly mixed with epinephrine. J Am Acad Dermatol. 2006 Jan;54(1):128-31. doi: 10.1016/j.jaad.2005.06.043. PMID 16384767
- [Background] Corah NL, Gale EN, Illig SJ. Assessment of a dental anxiety scale. J Am Dent Assoc. 1978 Nov;97(5):816-9. doi: 10.14219/jada.archive.1978.0394. PMID 31377
- [Background] Newton JT, Buck DJ. Anxiety and pain measures in dentistry: a guide to their quality and application. J Am Dent Assoc. 2000 Oct;131(10):1449-57. doi: 10.14219/jada.archive.2000.0056. PMID 11042984
- [Background] Heft MW, Parker SR. An experimental basis for revising the graphic rating scale for pain. Pain. 1984 Jun;19(2):153-61. doi: 10.1016/0304-3959(84)90835-2. PMID 6462727
- [Background] Whitcomb M, Drum M, Reader A, Nusstein J, Beck M. A prospective, randomized, double-blind study of the anesthetic efficacy of sodium bicarbonate buffered 2% lidocaine with 1:100,000 epinephrine in inferior alveolar nerve blocks. Anesth Prog. 2010 Summer;57(2):59-66. doi: 10.2344/0003-3006-57.2.59. PMID 20553136
- [Background] Corah NL. Development of a dental anxiety scale. J Dent Res. 1969 Jul-Aug;48(4):596. doi: 10.1177/00220345690480041801. No abstract available. PMID 5256508
- [Background] Catchlove RF. The influence of CO 2 and pH on local anesthetic action. J Pharmacol Exp Ther. 1972 May;181(2):298-309. No abstract available. PMID 4537424
- [Background] Ackerman WE 3rd, Ware TR, Juneja M. The air-liquid interface and the pH and PCO2 of alkalinized local anaesthetic solutions. Can J Anaesth. 1992 Apr;39(4):387-9. doi: 10.1007/BF03009051. PMID 1314142
- [Background] Benzon HT, Toleikis JR, Dixit P, Goodman I, Hill JA. Onset, intensity of blockade and somatosensory evoked potential changes of the lumbosacral dermatomes after epidural anesthesia with alkalinized lidocaine. Anesth Analg. 1993 Feb;76(2):328-32. PMID 8424510
- [Background] DiFazio CA, Carron H, Grosslight KR, Moscicki JC, Bolding WR, Johns RA. Comparison of pH-adjusted lidocaine solutions for epidural anesthesia. Anesth Analg. 1986 Jul;65(7):760-4. PMID 3717616

RESULTS

PARTICIPANT FLOW:
Groups:
- Buffered Lidocaine: administration of 4% buffered lidocaine with 1:100,000 epinephrine
  4% buffered lidocaine with 1:100,000 epinephrine
- Nonbuffered Lidocaine: administration of 4% lidocaine with 1:100,000 epinephrine
  4% lidocaine with 1:100,000 epinephrine
Period: Overall Study
Arm/Group | Buffered Lidocaine | Nonbuffered Lidocaine
Started | 45 | 43
Completed | 45 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buffered Lidocaine | Nonbuffered Lidocaine | Total
Number analyzed (Participants) | 45 | 43 | 88
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 43 | 88
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (13.0) | 36.3 (13.4) | 36.55 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 26 | 24 | 50
Region of Enrollment [Number; unit: participants]
  United States | 45 | 43 | 88

OUTCOME MEASURES:

1. Primary Outcome: Pain Measurement as Assessed on a Heft-Parker 170 mm Visual Analog Scale
Description: Patients will rate pain on a Heft-Parker visual analog scale during needle insertion, placement, and solution deposition phases of the anesthetic injection(s). Patients will also rate pain during the incision and dissection phases of the incision and drainage procedure. The number of millimeters along the scale are reported. No pain corresponded to 0 mm. Mild pain was defined as greater than 0 mm and less than or equal to 54 mm. Mild pain included the descriptors of "faint", "weak", and "mild pain". Moderate pain was defined as greater than 54 mm and less than 114 mm and included the descriptor "moderate". Severe pain was defined as equal to or greater than 114 mm up to and including 170 mm. Severe pain included the descriptors of "strong", "intense", and "maximum possible."
Time Frame: during incision/drainage on Day 0
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buffered Lidocaine | Nonbuffered Lidocaine
Number analyzed (Participants) | 45 | 43
units on a scale | 69.3 (60.1) | 59.2 (50.5)

2. Secondary Outcome: Postoperative Satisfaction on a 100 mm Visual Analog Scale
Description: Patients will rate their level of satisfaction with the incision and drainage procedure using a visual analog scale. The scale ranges from "not satisfied," to "somewhat satisfied," to "moderately satisfied," to "completely satisfied." Not satisfied corresponded to 0 mm. Somewhat satisfied was defined as greater than 0 mm and less than or equal to 33 mm. Moderately satisfied was defined as greater than 33 mm and less than 66 mm. Completely satisfied was defined as equal to or greater than 66 mm. Measurements along the scale were collected and analyzed by randomization test.
Time Frame: immediately post-procedure on Day 0
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buffered Lidocaine | Nonbuffered Lidocaine
Number analyzed (Participants) | 45 | 43
units on a scale | 92.7 (15.1) | 89.5 (13.7)

ADVERSE EVENTS:
Time Frame: Monitored and assessed during procedure on Day 0
Arm/Group | Buffered Lidocaine | Nonbuffered Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/43
Other Adverse Events (participants affected / at risk) | 0/45 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes